CLINICAL TRIAL: NCT02847520
Title: Validation of a Tool for Assessing Gambling Problems Related to the Practice of Poker: the Copenhagen Poker Screen (CHAPS)
Acronym: CHAPS
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC15_0054
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2016-07-28 (Estimated); Status verified 2016-07

CONDITIONS: Addiction
Keywords: Disorders related to gaming and gambling; poker
MeSH Terms: conditions — Behavior, Addictive; Gambling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Canadian Index Excessive Game — self-administered questionnaire Canadian Index Excessive Game

SUMMARY:
If the addiction to games of chance and gambling is a disease of increasing knowledge, the emergence of poker rout evaluation procedures, prevention and treatment usually offered to players in need. In the case of poker, which unlike other games has a real part to address and which damages are expressed differently, the evaluation can not be done identically to other games. This problem has often been emphasized in the literature, in particular the lack of specific tools for the identification of poker gambling problems. Thus, the fact of developing a specific evaluation tool could allow poker to take into account the specificity of poker among other games. This would be part of the evaluation complement batteries currently available to players in general by offering a specific tool, and secondly to allow the assessment of the aspects of the problems often absent for other games . The goal here is to develop and validate a specific tool detection of problem gambling in the particular context of poker.

ELIGIBILITY:
Inclusion Criteria:

* All subjects who had a practice of poker over the past 12 months

Exclusion Criteria:

* Participants who have already completed the survey (on the basis of their declaration)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Poker players
Sampling Method: Non-Probability Sample
Enrollment: 729 (Actual)
Dates: Start 2015-02; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
validate an evaluation tool of problem gambling within the specific framework of poker | 10 min

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Nantes, Nantes, France